CLINICAL TRIAL: NCT05328102
Title: A Phase 2 Randomized, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of XmAb13676 (Plamotamab) Combined With Tafasitamab Plus Lenalidomide Versus Tafasitamab Plus Lenalidomide in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Phase 2 Study of Plamotamab Combined With Tafasitamab Plus Lenalidomide Versus Tafasitamab Plus Lenalidomide in Relapsed or Refractory (R/R) Diffuse Large-cell B-cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated early by the sponsor due to business decision.
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb13676-03
Record Dates: First submitted 2022-04-04; First posted 2022-04-14 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large-cell B-cell Lymphoma
Keywords: DLBCL, NOS; Diffuse Large B-cell Lymphoma; Transformed indolent Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Part 1 Single Arm Multiple Dose Followed by Part 2 Randomized
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A: Plamotamab (lower dose), Tafasitamab, and Lenalidomide (Experimental): Drug: Plamotamab will be administered at a lower dose in addition to tafasitamab (12 milligrams [mg]/kilograms [kg] intravenously) plus lenalidomide (25 mg orally). This cohort was planned to enroll sequentially prior to Part 1B.
  Interventions: Biological: Plamotamab; Biological: Tafasitamab; Drug: Lenalidomide
- Part 1B: Plamotamab (target dose), Tafasitamab, and Lenalidomide (Experimental): Drug: Plamotamab will be administered at the target dose in addition to tafasitamab (12 mg/kg intravenously) plus lenalidomide (25 mg orally). This cohort was planned to enroll sequentially after Part 1A.
  Interventions: Biological: Plamotamab; Biological: Tafasitamab; Drug: Lenalidomide
- Part 2A :Plamotamab, Tafasitamab, and Lenalidomide (Experimental): Drug: Plamotamab will be administered at protocol defined dose in addition to tafasitamab (12 mg/kg intravenously) plus lenalidomide 25 mg (orally).
  Interventions: Biological: Plamotamab; Biological: Tafasitamab; Drug: Lenalidomide
- Part 2B: Tafasitamab and Lenalidomide (Active Comparator): Drug: Tafasitamab (12 mg/kg intravenously) plus lenalidomide 25 mg (orally).
  Interventions: Biological: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Plamotamab — Biological
  Other Names: XmAb13676
  Arms: Part 1A: Plamotamab (lower dose), Tafasitamab, and Lenalidomide; Part 1B: Plamotamab (target dose), Tafasitamab, and Lenalidomide; Part 2A :Plamotamab, Tafasitamab, and Lenalidomide
Biological: Tafasitamab — Biological
Drug: Lenalidomide — Drug

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of plamotamab when it is given with tafasitamab and lenalidomide in participants with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
This is a randomized, multicenter, open-label, Phase 2 study of plamotamab combined with tafasitamab plus lenalidomide versus tafasitamab plus lenalidomide in adult participants with DLBCL who have relapsed after or are refractory to at least 1 prior line of therapy, which must have included multi-agent chemoimmunotherapy inclusive of an anti-cluster of differentiation (CD) 20 monoclonal antibody, and who are not candidates for autologous stem-cell transplantation (ASCT), refuse ASCT, or relapse after ASCT.

The study was planned to be performed sequentially, with Part 1A (Safety run-in, with a lower plamotamab dose), Part 1B (Safety run-in, with the target plamotamab dose) and Part 2 (Open-Label, randomized). The study was terminated by the Sponsor during Part 1A of the study. No participants were enrolled in Part 1B or Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of DLBCL, not otherwise specified, including DLBCL arising from low grade lymphoma
* CD20+ and CD19+ lymphoma
* Archival paraffin embedded tumor tissue or unstained slides must be available for retrospective cell of origin determination
* Relapsed or refractory
* At least 1 prior systemic line(s) of therapy, one of which must have included multi-agent chemoimmunotherapy that includes an anti-CD20 monoclonal antibody.
* At least 1 bidimensionally measurable disease site. The lesion must have a greatest transverse diameter of ≥ 1.5 centimeter (cm) and greatest perpendicular diameter of ≥ 1.0 cm at baseline. The lesion must have a positive finding on positron emission tomography (PET) scan
* Ineligible for or refuse hematopoietic stem cell transplantation (HSCT).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Completed vaccination for the SARS-CoV-2 virus prior to study entry
* Fertile participants must agree to use 2 highly effective methods of birth control during for at least 6 months (male participants) and 8 months (female participants) after the last dose of study treatment

Exclusion Criteria:

* Any other histological type of lymphoma, including high-grade B-cell lymphoma, including those with myelocytomatosis oncogene (MYC) and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements primary mediastinal (thymic) large B cell (PMBL) or Burkitt lymphoma
* A prior diagnosis of chronic lymphocytic leukemia (CLL) (Richter's Transformation)
* Primary central nervous system lymphoma

Exclusionary Previous and Current Treatment:

* Previously received treatment with an anti-CD20 × anti-CD3 bispecific antibody (bsAb)
* Anti-CD20 therapy (for example, rituximab) within 21 days prior to study entry
* Participants who have, within 14 days prior study entry:

  * Chemotherapy, radiotherapy, or other lymphoma-specific therapy not including anti CD20 therapy
  * Small molecule or investigational anticancer agents within 6 elimination half-lives
  * Received live vaccines within 30 days
  * Required systemic anti-infective therapy for active, intercurrent infections
* Participants who have had the following prior therapies or treatments:

  * Were previously treated with CD19-targeted therapy, including chimeric antigen receptor-T cell (CAR-T), unless current biopsy is CD19+
  * Have a history of hypersensitivity to compounds of similar biological or chemical composition to tafasitamab, immunomodulatory imide drugs (IMiDs)
  * Previous allogenic stem cell transplantation
  * Have a history of deep venous thrombosis/embolism, threatening thromboembolism
  * Concurrently use other anticancer or experimental treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chiarella, Study Director — Senior Director, Clinical Science, Clinical Development
Locations (3):
- Swedish Cancer Center, Seattle, Washington, United States
- CHU de Rennes - Hopital de Pontchaillou, Rennes, France
- Hospital Universitario Virgen de las Nieves, Granada, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned to enroll participants at 11 sites (1 in the United States, 7 in France, 2 in Spain, and 1 in South Korea). However, due to early study termination only 3 participants were enrolled and dosed at a single site in the United States.
Pre-assignment Details: The study was planned to be performed sequentially, with Part 1A (Safety run-in, with a lower plamotamab dose), Part 1B (Safety run-in, with the target plamotamab dose) and Part 2 (Open-Label, randomized). The study was terminated by the Sponsor during Part 1A of the study. No participants were enrolled in Part 1B or Part 2.
Groups:
- Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide: Plamotamab was administered at a lower dose in addition to tafasitamab (12 milligrams [mg]/kilograms [kg] intravenously) plus lenalidomide (25 mg orally).
Period: Overall Study
Arm/Group | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide
Started | 3
Received at Least 1 Dose of Study Drug | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Enrolled Analysis Set: All participants who signed the informed consent form, were determined to be eligible, and received Day -8 tafasitamab dose (Study Day 1). The study was terminated by the Sponsor during Part 1A of the study. No participants were enrolled in Part 1B or Part 2.
Groups:
- Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide: Plamotamab was administered at a lower dose in addition to tafasitamab (12 mg/kg intravenously) plus lenalidomide (25 mg orally).
Arm/Group | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.

OUTCOME MEASURES:

1. Primary Outcome: Part 1 A: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant. The AE did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug. AEs may have included the onset of new illness and the exacerbation of preexisting conditions. TEAEs were defined as events with onset dates on or after the start of study treatment or events that were present before the first infusion of study treatment and subsequently worsened in severity. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From first dose of study drug up to end of treatment (maximum treatment exposure: 303 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Part 1 A: Number of Participants With Cytokine Release Syndrome
Description: Cytokine release syndrome was defined as "a supraphysiologic response following any immune therapy that results in the activation or engagement of endogenous or infused T cells and/or other immune effector cells". A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From first dose of study drug up to end of treatment (maximum treatment exposure: 303 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of treatment (maximum treatment exposure: 303 days)
Description: Enrolled Analysis Set: All participants who signed the informed consent form, were determined to be eligible, and received Day -8 tafasitamab dose (Study Day 1). The study was terminated by the Sponsor during Part 1A of the study. No participants were enrolled in Part 1B or Part 2.
Arm/Group | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide (N=3)
Cytokine release syndrome (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Pneumonia aspiration (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Volvulus of small bowel (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: Plamotamab (Lower Dose), Tafasitamab, and Lenalidomide (N=3)
Cytokine release syndrome (Immune system disorders) | 2
Fatigue (General disorders) | 2
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Oedema peripheral (General disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Blood creatinine increased (Investigations) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Pyrexia (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Asthenia (General disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Embolism (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study in Part 1A, only 3 participants enrolled. No participants were enrolled in Part 1B or Part 2. Safety data is limited due to the small sample size. No efficacy data was collected for the secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05328102/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT05328102/SAP_001.pdf